CLINICAL TRIAL: NCT01695525
Title: Neurocardiogenic Syncope and the Role That Yoga Plays in People With Autonomic Dysfunction
Brief Title: Influence of Yoga in Patients With Neurocardiogenic Syncope
Acronym: SYNC - YOGA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dhanunjaya Lakkireddy, MD, FACC (Other)
Responsible Party: Sponsor-Investigator, Dhanunjaya Lakkireddy, MD, FACC, Professor of Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12945
Record Dates: First submitted 2012-07-05; First posted 2012-09-28 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Syncope, Vasovagal
Keywords: Neurocardiogenic Syncope; Yoga
MeSH Terms: conditions — Syncope, Vasovagal | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga (Experimental): Participants will be asked to practice Yoga 3 times per week at a minimum, and daily at a maximum. Participants will receive training in different Yoga techniques including breathing exercises, postures and meditation. Participants will be asked to practice 1 hour Yoga sessions comprised of breathing exercises, postures and meditation.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — Includes breathing exercises, postures, and meditation. Participant practices yoga at their home a minimum of 3 times per week for 1 hour per time. Participation can last for up to 1 year.

SUMMARY:
Syncope is a common problem that many clinicians may encounter in various outpatient settings. Neurocardiogenic syncope (NCS) is a benign condition characterized by a self limited episode of systemic hypotension. Patients are usually managed with education on syncope, anxiety management, and coping skills.

It has been established that practice of Yoga could relieve stress and anxiety. In a different study, they also found that Yoga positively influences cardiovascular function by decreasing the heart rate and blood pressure. The main objective of Yoga is to achieve control over the autonomic nervous system and able to control functions like heart rate, blood pressure and respiratory rate.

Based on the findings that Yoga relieves stress and reduces heart rate, the investigators propose to study if Yoga can decrease the frequency of NCS and also reduce the symptoms associated with these episodes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent Neurocardiogenic syncope
* At least one episode of syncope or pre-syncopal event in the last 3 months prior to enrollment

Exclusion Criteria:

* Previously established diagnosis of any psychiatric illness.
* Previous history of Coronary Artery Disease, myocardial infarction, congestive heart failure, carotid sinus hypersensitivity
* Established diagnosis of tachy and/or brady arrhythmias, except cardioinhibiotry neurocardiogenic syncope.
* History of pacemaker, ICD or CRT-D implantation.
* Other conditions where Yoga should be avoided are:

  1. Pregnant women
  2. Subjects with untreated or uncontrolled high blood pressure
  3. Subjects with past history of Pnuemothorax.
  4. Subjects with severe cervical spondylitis and cervical, thoracic or lumbar disc prolapse.
  5. Subjects with carotid stenosis
  6. Subjects with history of psychosis (evidence of acute episodes with deep and prolonged meditation) or substance abuse.
  7. Subjects with the history of epilepsy ( evidence of acute episodes with deep and prolonged meditation)
  8. Subjects with glaucoma
  9. Subjects with history of Total Hip Replacement.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in frequency of recurrent syncopal spells in patients with Neurocardiogenic syncope (NCS) | Baseline to 3 Months
  Differences in the incidence of syncopal spells pre and post Yoga.
Change in frequency of recurrent syncopal spells in patients with Neurocardiogenic syncope (NCS) | Baseline to 1 Year
  Differences in the incidence of syncopal spells pre and post Yoga.
Change in frequency of recurrent syncopal spells in patients with Neurocardiogenic syncope (NCS) | Baseline to 1 Year
  Differences in the incidence of syncopal symptoms pre and post Yoga.

SECONDARY OUTCOMES:
Change in Heart Health | 3 Months, 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, FACC, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States